CLINICAL TRIAL: NCT02913508
Title: A Randomized, Open Label Phase 2 Study to Assess Pharmacokinetics, Pharmacodynamics, Immunogenicity, Safety and Exploratory Efficacy of Vedolizumab Subcutaneous Compared to Vedolizumab Intravenous in Subjects With Moderately to Severely Active Ulcerative Colitis or Crohn's Disease
Brief Title: Vedolizumab Subcutaneous (SC) Versus Intravenous (IV) in Ulcerative Colitis or Crohn's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLN0002SC_201; 2013-003030-32 (EudraCT Number); U1111-1146-5451 (Other: WHO (UTN))
Record Dates: First submitted 2016-09-22; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Vedolizumab 300 mg IV Q8W (Experimental): Vedolizumab 300 mg, intravenously, at Weeks 0 and 2, and then every 8 weeks (Q8W) (Weeks 6 and 14).
  Interventions: Drug: Vedolizumab intravenous injection
- Vedolizumab 300 mg IV / 160 mg SC Q3W (Experimental): Vedolizumab 300 mg, intravenously, at Weeks 0 and 2, then vedolizumab 160 mg, subcutaneously (SC), every 3 weeks (Q3W) (Weeks 6, 9, 12, 15 and 18).
  Interventions: Drug: Vedolizumab intravenous injection; Drug: Vedolizumab subcutaneous injection
- Vedolizumab 300 mg IV / 108 mg SC Q2W (Experimental): Vedolizumab 300 mg, intravenously, at Weeks 0 and 2, then vedolizumab 108 mg, subcutaneously, every 2 weeks (Q2W) (Weeks 6, 8, 10, 12, 14, 16, 18 and 20).
  Interventions: Drug: Vedolizumab intravenous injection; Drug: Vedolizumab subcutaneous injection
- Vedolizumab 480 mg SC / 160 mg SC Q3W (Experimental): Vedolizumab 480 mg, subcutaneously, at Weeks 0 and 2, then vedolizumab 160 mg, subcutaneously, every 3 weeks (Weeks 6, 9, 12, 15 and 18).
  Interventions: Drug: Vedolizumab subcutaneous injection
- Vedolizumab 324 mg SC / 108 mg SC Q2W (Experimental): Vedolizumab 324 mg, subcutaneously, at Weeks 0 and 2, then vedolizumab 108 mg, subcutaneously, every 2 weeks (Weeks 6, 8, 10, 12, 14, 16, 18 and 20).
  Interventions: Drug: Vedolizumab subcutaneous injection

INTERVENTIONS:
Drug: Vedolizumab intravenous injection — Vedolizumab intravenous injection
  Other Names: MLN0002; Entyvio
  Arms: Vedolizumab 300 mg IV / 108 mg SC Q2W; Vedolizumab 300 mg IV / 160 mg SC Q3W; Vedolizumab 300 mg IV Q8W
Drug: Vedolizumab subcutaneous injection — Vedolizumab subcutaneous injection
  Other Names: MLN0002SC
  Arms: Vedolizumab 300 mg IV / 108 mg SC Q2W; Vedolizumab 300 mg IV / 160 mg SC Q3W; Vedolizumab 324 mg SC / 108 mg SC Q2W; Vedolizumab 480 mg SC / 160 mg SC Q3W

SUMMARY:
The purpose of this study is to assess the bioavailability and pharmacokinetics (PK) of multiple doses of vedolizumab subcutaneous (SC) compared to vedolizumab intravenous (IV).

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to determine its availability and reaction in the body of people who have moderately to severely active Ulcerative Colitis (UC) or Crohn's Disease (CD). This study will look at the availability and reaction of vedolizumab in people who are administered the treatment subcutaneously (SC) compared people who are administered the treatment intravenously (IV).

The study will enroll approximately 200 patients with moderately to severely active UC or CD. Participants will be randomly assigned (by chance, like flipping a coin) to one of the five treatment groups:

* vedolizumab 300 mg IV
* vedolizumab 300 mg IV and vedolizumab 160 mg SC
* vedolizumab 300 mg IV and vedolizumab 108 mg SC
* vedolizumab 480 mg SC and vedolizumab 160 mg SC
* vedolizumab 324 mg SC and vedolizumab 108 mg SC

All participants will receive one of the treatments they are assigned to at various treatment visits throughout the study.

This multi-centre trial will be conducted in North America, Europe and Asia. The overall time to participate in this study is approximately 41 weeks in addition to a follow-up survey that will be administered every 6 months for 2 years. Participants will make 16 visits to the clinic, including a safety follow-up assessment 18 weeks after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedure.
3. Is aged 18 to 80 years, inclusive.
4. The male or female participant is voluntarily able to give informed consent.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.
6. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.

   Inclusion Criteria for Ulcerative Colitis Participants
7. Has a diagnosis of ulcerative colitis (UC) established at least 3 months prior to randomization by clinical and endoscopic evidence and corroborated by a histopathology report.
8. Has moderately to severely active UC as determined by a partial Mayo score of 3 to 9 within 7 days prior to the first dose of study drug.
9. Has evidence of UC extending proximal to the rectum (≥15 cm of involved colon).
10. Participants with extensive colitis or pancolitis of >8 years duration or left-sided colitis of >12 years duration must have documented evidence that a surveillance colonoscopy with random and targeted biopsies was performed within 18 months of the initial screening visit (may be performed during screening).
11. Participants with a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factor for colorectal cancer must be up-to-date on colorectal cancer surveillance (may be performed during screening).
12. Participants may be receiving a therapeutic dose of the following drugs:

    1. Oral or topical (rectal) 5-aminosalicylate (5-ASA) compounds provided that the dose has been stable for the 2 weeks immediately prior to randomization;
    2. Oral corticosteroid therapy (prednisone at a stable dose ≤30 mg/day, budesonide at a dose ≤9 mg/day or equivalent steroid) provided that the dose has been stable for the 4 weeks immediately prior to randomization if corticosteroids have just been initiated, or for the 2 weeks immediately prior to randomization if corticosteroids are being tapered;
    3. Topical (rectal) corticosteroid enemas/suppositories;
    4. Azathioprine or 6-mercaptopurin provided that the dose has been stable for the 8 weeks immediately prior to randomization;
    5. Antidiarrheals (eg, loperamide, diphenoxylate with atropine) for control of chronic diarrhea;
    6. Probiotics (eg, Culturelle, S. boulardii) provided that the dose has been stable for the 2 weeks immediately prior to randomization;
    7. Antibiotics used for the treatment of inflammatory bowel disease (IBD) (ie, ciprofloxacin, metronidazole).

    Inclusion Criteria for Crohn's Disease Participants
13. Has a diagnosis of Crohn's Disease (CD) established at least 3 months prior to randomization by clinical and endoscopic evidence and corroborated by a histopathology report. Cases of CD established at least 3 months prior to randomization for which a histopathology report is not available will be considered based on the weight of the evidence supporting the diagnosis and excluding other potential diagnoses, and must be discussed with the sponsor on a case-by-case basis prior to randomization.
14. Has moderately to severely active CD as determined by Crohn's Disease Activity Index (CDAI) score of 220 to 450 within 7 days prior to the first dose of study drug and 1 of the following:

    1. C-reactive protein (CRP) level >2.87 mg/L during the Screening Period, OR;
    2. Ileocolonoscopy with photographic documentation of a minimum of 3 nonanastomotic ulcerations (each >0.5 cm in diameter) or 10 aphthous ulcerations (involving a minimum of 10 contiguous cm of intestine) consistent with CD, within 4 months prior to randomization, OR;
    3. Fecal calprotectin >250 mcg/g stool during the Screening Period in conjunction with Computed Tomography (CT) enterography, magnetic resonance (MR) enterography, contrast-enhanced small bowel radiography, or wireless capsule endoscopy revealing Crohn's ulcerations (aphthae not sufficient), within 4 months prior to screening (participants with evidence of fixed stenosis or small bowel stenosis with prestenotic dilation should not be included).
15. Has CD involvement of the ileum and/or colon, at a minimum.
16. Participants with extensive colitis or pancolitis of >8 years duration or limited colitis of >12 years duration must have documented evidence that a surveillance colonoscopy with random and targeted biopsies was performed within 18 months of randomization (may be performed during screening).
17. Participants with a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factor for colorectal cancer must be up-to-date on colorectal cancer surveillance (may be performed during screening).
18. Participants may be receiving a therapeutic dose of the following drugs:

    1. Oral or topical (rectal) 5-ASA compounds provided that the dose has been stable for the 2 weeks immediately prior to randomization;
    2. Oral corticosteroid therapy (prednisone at a stable dose ≤30 mg/day, budesonide at a dose ≤9 mg/day, or equivalent steroid) provided that the dose has been stable for the 4 weeks immediately prior to randomization if corticosteroids have just been initiated, or for the 2 weeks immediately prior to randomization if corticosteroids are being tapered;
    3. Topical (rectal) corticosteroid enemas/suppositories;
    4. Antibiotics used for the treatment of IBD (ie, ciprofloxacin, metronidazole);
    5. Azathioprine or 6-mercaptopurin provided that the dose has been stable for the 8 weeks immediately prior to randomization;
    6. Methotrexate provided that the dose has been stable for the 8 weeks immediately prior to randomization;
    7. Antidiarrheals (eg, loperamide, diphenoxylate with atropine) for control of chronic diarrhea;
    8. Probiotics (eg, Culturelle, S. boulardii) provided that the dose has been stable for the 2 weeks immediately prior to randomization.

Exclusion Criteria

Gastrointestinal Exclusion Criteria:

1. Evidence of abdominal abscess at the initial Screening Visit.
2. Extensive colonic resection, subtotal or total colectomy.
3. History of >3 small bowel resections or diagnosis of short bowel syndrome.
4. Have received tube feeding, defined formula diets, or parenteral alimentation within 21 days prior to the administration of the first dose of study drug.
5. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
6. Within 30 days prior to randomization, have received any of the following for the treatment of underlying disease: a) Any investigational or approved nonbiologic therapy for UC or CD (eg, cyclosporine, thalidomide) other than those specified in the protocol.
7. Within 60 days prior to randomization, have received any of the following:

   1. Infliximab,
   2. Certolizumabpegol,
   3. Adalimumab,
   4. Golimumab,
   5. Any other investigational or approved biological agent, other than local injections for non IBD conditions (eg, intra-ocular injections for the treatment of wet macular degeneration).
8. Evidence of or treatment for clostridium difficile infection or other intestinal pathogen within 28 days prior to randomization.
9. Currently require or are anticipated to require major surgical intervention during the study.
10. History or evidence of adenomatous colonic polyps that have not been removed.
11. History or evidence of colonic mucosal dysplasia.

    Infectious Disease Exclusion Criteria
12. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), or a known history of human immunodeficiency virus infection (HIV) at Screening.
13. Active or latent tuberculosis (TB), regardless of treatment history, as evidenced by any of the following:

    1. History of TB,
    2. A positive diagnostic TB test within 1 month of randomization defined as:

    i. a positive QuantiFERON® test or 2 successive indeterminate QuantiFERON® tests, OR ii. a tuberculin skin test reaction ≥10 mm (≥5 mm in participants receiving the equivalent of >15 mg/day prednisone), c. Chest X-ray within 3 months of randomization in which active or latent pulmonary tuberculosis cannot be excluded.
14. Any identified congenital or acquired immunodeficiency (eg, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
15. Any live vaccinations within 30 days prior to study drug administration except for the influenza vaccine.
16. Clinically significant extra-intestinal infection (eg, pneumonia, pyelonephritis) or abdominal abscess within 30 days of the initial Screening visit.

    General Exclusion Criteria
17. Previous exposure to vedolizumab.
18. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
19. Has a positive test for drug screening.
20. Any prior exposure to natalizumab, efalizumab, or rituximab.
21. Female participants who are lactating or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 prior to study drug administration.
22. Any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise participant's safety.
23. Had any surgical procedure requiring general anesthesia within 30 days prior to randomization or is planning to undergo major surgery during the study period.
24. Any history of malignancy, except for the following:

    1. adequately-treated nonmetastatic basal cell skin cancer;
    2. squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to randomization; and
    3. history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to randomization. Participants with remote history of malignancy (eg, >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis prior to randomization.
25. History of any major neurological disorders, including but not limited to stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
26. Positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist prior to the administration of the first dose of study drug.
27. Any of the following laboratory abnormalities during the Screening period:

    1. Hemoglobin level <8 g/dL,
    2. White blood cell (WBC) count <3 x 10^9/L,
    3. Lymphocyte count <0.5 x 10^9/L,
    4. Platelet count <100 x 10^9/L or >1200 x10^9/L,
    5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 x the upper limit of normal (ULN),
    6. Alkalinephosphatase>3xULN,
    7. Serum creatinine >2 x ULN,
    8. Albumin <2.0 g/dL (<20 g/L).
28. Current or recent history (within 1 year prior to randomization) of alcohol dependence or illicit drug use.
29. Active psychiatric problems that, in the investigator's opinion, may interfere with compliance with the study procedures.
30. Unable to attend all the study visits or comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Average Concentration of Vedolizumab Over the Dosing Interval at Steady-State (Cavg, ss) | Week 0 up to Week 22
  Cavg, ss is defined as the average concentration over the dosing interval at steady-state, calculated as area under the serum concentration-time curve over the dosing interval at steady-state(AUCss)/Tau, where Tau is the dosing interval.
Average Concentration of Vedolizumab Over the Dosing Interval from Week 0 to Week 6 (Cavg[wk0-6]) | Week 0 to Week 6
  Area under the serum concentration-time curve from Week 0 to Week 6, calculated using the linear trapezoidal rule.

SECONDARY OUTCOMES:
Percentage of Participants with Positive Human Antihuman Antibody (HAHA) During the Study | Pre-dose at Weeks 0, 2, 6, 10, 18, 22 and 38
Percentage of Participants with Positive Neutralizing Human Antihuman Antibody (HAHA) During the Study | Pre-dose at Weeks 0, 2, 6, 10, 18, 22 and 38
  Only participants with positive HAHA will be evaluated for positive neutralizing HAHA.
Percent Saturation of Mucosal Addressin Cell Adhesion Molecule-1 (MAdCAM-1) at Week 6 | Week 6
Percent Saturation of Mucosal Addressin Cell Adhesion Molecule-1 (MAdCAM-1) at Week 22 | Week 22

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda